CLINICAL TRIAL: NCT05885373
Title: A Single-arm, Open-label Clinical Study to Evaluate the Effect of SIM01 in Female Subjects With Non-Alcoholic Fatty Liver Disease (NAFLD)
Brief Title: A Clinical Study to Evaluate the Effect of SIM01 in Female With NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GenieBiome Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GB-NAFLD
Record Dates: First submitted 2023-04-14; First posted 2023-06-01 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Non-Alcoholic Fatty Liver Disease; Probiotics
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: All study subjects will receive the same study products.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIM01 (Experimental): 2 sachets daily for 3 months
  Interventions: Dietary Supplement: SIM01

INTERVENTIONS:
Dietary Supplement: SIM01 — SIM01 consists of a blend of food-grade Bifidobacterium as active probiotics
  Other Names: G-NiiB Immunity formula

SUMMARY:
Non-alcoholic fatty liver disease is one of the most common chronic liver diseases worldwide. Available data indicates that probiotics may regulate the gut microbiota and improve liver function in females with non-alcoholic fatty liver disease. In this study, we aim to investigate if the synbiotics (prebiotics and probiotics) are efficacious subjects in liver function improvement in female subjects with Non-alcoholic fatty liver disease.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is one of the most common chronic liver diseases worldwide.(1) The prevalence of NAFLD is estimated to be about 20%-30% in the Western world (2) and increasing in Asia. The prevalence of NAFLD across Asia varies from 5% to 40%.(3,4) In one study with a sample of 922 subjects using proton-magnetic resonance spectroscopy and transient elastography, 252 subjects had intrahepatic triglyceride content ≥5%, and the population prevalence of NAFLD in Hong Kong Chinese was 27.3%.1 NAFLD may progress to non-alcoholic steatohepatitis (NASH), cirrhosis, liver failure and liver cancer, and is believed to be the leading etiology for cryptogenic cirrhosis.(5,6) NAFLD is also strongly associated with obesity and metabolic syndrome and is shown to be an independent cardiovascular risk factor.(7,8)

At present, there is no standard pharmacologic therapy available for NAFLD currently. Current management for NAFLD includes diet and lifestyle changes, management of underlying metabolic risk factors and pharmacological therapies. Insulin-sensitizing medication such as Pioglitazone has been shown to improve histological NASH in terms of steatosis, inflammation, ballooning, NAFLD Activity Score (NAS score) and resolution of NASH. (9) However, the long-term efficacy and safety of Pioglitazone are unknown, and not all patients respond to Pioglitazone. Vitamin E is a fat-soluble compound which prevents liver injury by blocking intrinsic apoptotic pathways and by protecting against mitochondrial toxicity. (10) It also improves histological NASH in terms of steatosis, inflammation, ballooning, NAS score, and resolution of NASH at a dose of 800 IU/day. (9) However, the long-term safety of vitamin E is also an issue, because doses of 400 IU/day or higher have been associated with increased all-cause mortality. (11) While lifestyle management is often advocated, it is difficult to maintain. (12) Thus, it is important to explore new treatment strategies.

In general, NAFLD prevalence is higher in men compared to women. However, the prevalence of NAFLD in women is increasing in women over the past 10 years, (13) especially postmenopausal women who have greater NAFLD risk and higher rates of severe hepatic fibrosis relative to premenopausal women, and older women with NAFLD experience greater mortality than men. (14) A cohort study in Japan reported that women after the age of 70 had a higher prevalence of fatty liver than men (19.4% vs 14.9%). (15) Another cohort showed that gradual age-related increases in NAFLD prevalence were also observed in women (3.9% in the 21-39 age group; 7.6% in the 40-49 age group; 14.0% in the 50-59 age group; 18.9% in 60-69 age group), but not men. (15)

NAFLD is more prevalent in overweight and obese individuals; gut microbiota also plays a role in the development of insulin resistance, hepatic steatosis, necroinflammation and fibrosis. (16) On the other hand, probiotics can strengthen the intestinal wall, reducing its permeability, bacterial translocation, and endotoxemia according to animal and human studies. Recently, it has been reported that NAFLD might be linked to small intestinal bacterial overgrowth (SIBO), which induces liver injury by gut-derived lipopolysaccharides (LPS) and TNF- α production. (17) Probiotics have several anti-inflammatory effects that can contribute to their clinical benefits in NAFLD. (18)

The use of probiotics, prebiotics and synbiotics has been considered a potential and promising strategy to regulate the gut microbiota. (19, 20) Some clinical studies have been conducted to investigate the effects of probiotics on liver functions in NAFLD and NASH subjects. In general, the results of the trials (21-28) showed that the use of probiotics can reduce BMI, total fat percentage, total cholesterol, triglycerides, fasting insulin, alanine aminotransferase (ALT), aspartate transaminase (AST), tumour necrosis factor (TNF-α), interleukin (IL-6), liver stiffness et cetera.

This is a single-arm, open-label clinical trial for evaluating the efficacy of SIM01 on the reduction of liver biochemistry in 40 female subjects with NAFLD. All subjects will take 2 sachets of SIM01 daily for 3 months with monthly assessment on adverse event observation, and adherence to the study product throughout the study period. The change in CAP scores measured by the fibroscan, BMI, liver function and interleukin-6 will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects with NAFLD with CAP ≥ 270 by fibroscan
* Age ≥ 55
* Subjects with or without diabetes or components of metabolic syndrome and having stable medication 3 months prior to enrolment
* Written informed consent can be obtained

Exclusion Criteria:

* Known history of any secondary causes of NAFLD including alcoholic liver disease, drug-induced liver injury, autoimmune hepatitis, viral hepatitis, cholestatic liver disease and metabolic/genetic liver disease
* Known diabetes with poor control (HbA1c > 8.5%) within 3 months
* Significant alcohol consumption (over 10g per day: a half pint or half bottle of beer or a standard-size of a wine glass)
* Consumption of systemic corticosteroids or methotrexate in the last 6 months
* Concomitant probiotics or prebiotics one month prior to enrolment
* Any condition or allergy history for probiotics
* Subjects who are using antibiotics, insulin and Glucagon-like peptide-1(GLP1) such as dulaglutide, semaglutide
* Malignancy

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Controlled Attenuation Parameter (CAP) score by fibroscan after taking SIM01 for 3 months | 3 months
  The change of CAP score measured by fibroscan. CAP score is a measurement of fat accumulation in the liver to further determine the steatosis grade. The CAP score ranges from 100 to 400 decibels per meter (dB/m). The higher the score, the more the steatosis is.

SECONDARY OUTCOMES:
Change in liver enzymes (alanine aminotransferase (ALT) and aspartate transaminase (AST)) across the study period. | 3 months
  The change in the level of liver enzymes.
Change in fasting lipid and HbA1c across the study period. | 3 months
  The change in the level of lipid profiles
Change of body mass index (BMI) across the study period. | 3 months
  The change of body weight and body height
Change of body waist circumference across the study period. | 3 months
  The change of waist circumference
Change in interleukin-6 (IL-6) across the study period. | 3 months
  The change in the one of the immunity marker

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Ching, PhD, Study Director — GenieBiome Limited
Locations (1):
- GenieBiome Limited, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amarapurkar DN, Hashimoto E, Lesmana LA, Sollano JD, Chen PJ, Goh KL; Asia-Pacific Working Party on NAFLD. How common is non-alcoholic fatty liver disease in the Asia-Pacific region and are there local differences? J Gastroenterol Hepatol. 2007 Jun;22(6):788-93. doi: 10.1111/j.1440-1746.2007.05042.x. PMID 17565631
- [Background] Caldwell SH, Oelsner DH, Iezzoni JC, Hespenheide EE, Battle EH, Driscoll CJ. Cryptogenic cirrhosis: clinical characterization and risk factors for underlying disease. Hepatology. 1999 Mar;29(3):664-9. doi: 10.1002/hep.510290347. PMID 10051466
- [Background] Farrell GC, Larter CZ. Nonalcoholic fatty liver disease: from steatosis to cirrhosis. Hepatology. 2006 Feb;43(2 Suppl 1):S99-S112. doi: 10.1002/hep.20973. PMID 16447287
- [Background] Hamaguchi M, Kojima T, Takeda N, Nagata C, Takeda J, Sarui H, Kawahito Y, Yoshida N, Suetsugu A, Kato T, Okuda J, Ida K, Yoshikawa T. Nonalcoholic fatty liver disease is a novel predictor of cardiovascular disease. World J Gastroenterol. 2007 Mar 14;13(10):1579-84. doi: 10.3748/wjg.v13.i10.1579. PMID 17461452
- [Background] Wong VW, Wong GL, Yip GW, Lo AO, Limquiaco J, Chu WC, Chim AM, Yu CM, Yu J, Chan FK, Sung JJ, Chan HL. Coronary artery disease and cardiovascular outcomes in patients with non-alcoholic fatty liver disease. Gut. 2011 Dec;60(12):1721-7. doi: 10.1136/gut.2011.242016. Epub 2011 May 20. PMID 21602530
- [Background] Wong VW, Chu WC, Wong GL, Chan RS, Chim AM, Ong A, Yeung DK, Yiu KK, Chu SH, Woo J, Chan FK, Chan HL. Prevalence of non-alcoholic fatty liver disease and advanced fibrosis in Hong Kong Chinese: a population study using proton-magnetic resonance spectroscopy and transient elastography. Gut. 2012 Mar;61(3):409-15. doi: 10.1136/gutjnl-2011-300342. Epub 2011 Aug 16. PMID 21846782
- [Background] Bellentani S, Scaglioni F, Marino M, Bedogni G. Epidemiology of non-alcoholic fatty liver disease. Dig Dis. 2010;28(1):155-61. doi: 10.1159/000282080. Epub 2010 May 7. PMID 20460905
- [Background] Chitturi S, Wong VW, Farrell G. Nonalcoholic fatty liver in Asia: Firmly entrenched and rapidly gaining ground. J Gastroenterol Hepatol. 2011 Jan;26 Suppl 1:163-72. doi: 10.1111/j.1440-1746.2010.06548.x. PMID 21199528
- [Background] Sanyal AJ, Chalasani N, Kowdley KV, McCullough A, Diehl AM, Bass NM, Neuschwander-Tetri BA, Lavine JE, Tonascia J, Unalp A, Van Natta M, Clark J, Brunt EM, Kleiner DE, Hoofnagle JH, Robuck PR; NASH CRN. Pioglitazone, vitamin E, or placebo for nonalcoholic steatohepatitis. N Engl J Med. 2010 May 6;362(18):1675-85. doi: 10.1056/NEJMoa0907929. Epub 2010 Apr 28. PMID 20427778
- [Background] Soden JS, Devereaux MW, Haas JE, Gumpricht E, Dahl R, Gralla J, Traber MG, Sokol RJ. Subcutaneous vitamin E ameliorates liver injury in an in vivo model of steatocholestasis. Hepatology. 2007 Aug;46(2):485-95. doi: 10.1002/hep.21690. PMID 17659596
- [Background] Miller ER 3rd, Pastor-Barriuso R, Dalal D, Riemersma RA, Appel LJ, Guallar E. Meta-analysis: high-dosage vitamin E supplementation may increase all-cause mortality. Ann Intern Med. 2005 Jan 4;142(1):37-46. doi: 10.7326/0003-4819-142-1-200501040-00110. Epub 2004 Nov 10. PMID 15537682
- [Background] Rodriguez-Hernandez H, Cervantes-Huerta M, Rodriguez-Moran M, Guerrero-Romero F. Decrease of aminotransferase levels in obese women is related to body weight reduction, irrespective of type of diet. Ann Hepatol. 2011 Oct-Dec;10(4):486-92. PMID 21911890
- [Background] Arshad T, Golabi P, Paik J, Mishra A, Younossi ZM. Prevalence of Nonalcoholic Fatty Liver Disease in the Female Population. Hepatol Commun. 2018 Nov 27;3(1):74-83. doi: 10.1002/hep4.1285. eCollection 2019 Jan. PMID 30619996
- [Background] DiStefano JK. NAFLD and NASH in Postmenopausal Women: Implications for Diagnosis and Treatment. Endocrinology. 2020 Oct 1;161(10):bqaa134. doi: 10.1210/endocr/bqaa134. PMID 32776116
- [Background] Hamaguchi M, Kojima T, Ohbora A, Takeda N, Fukui M, Kato T. Aging is a risk factor of nonalcoholic fatty liver disease in premenopausal women. World J Gastroenterol. 2012 Jan 21;18(3):237-43. doi: 10.3748/wjg.v18.i3.237. PMID 22294826
- [Background] Eslamparast T, Eghtesad S, Hekmatdoost A, Poustchi H. Probiotics and Nonalcoholic Fatty liver Disease. Middle East J Dig Dis. 2013 Jul;5(3):129-36. PMID 24829682
- [Background] Loguercio C, De Simone T, Federico A, Terracciano F, Tuccillo C, Di Chicco M, Carteni M. Gut-liver axis: a new point of attack to treat chronic liver damage? Am J Gastroenterol. 2002 Aug;97(8):2144-6. doi: 10.1111/j.1572-0241.2002.05942.x. No abstract available. PMID 12190198
- [Background] Solga SF, Diehl AM. Non-alcoholic fatty liver disease: lumen-liver interactions and possible role for probiotics. J Hepatol. 2003 May;38(5):681-7. doi: 10.1016/s0168-8278(03)00097-7. No abstract available. PMID 12713883
- [Background] Pandey KR, Naik SR, Vakil BV. Probiotics, prebiotics and synbiotics- a review. J Food Sci Technol. 2015 Dec;52(12):7577-87. doi: 10.1007/s13197-015-1921-1. Epub 2015 Jul 22. PMID 26604335
- [Background] Yadav MK, Kumari I, Singh B, Sharma KK, Tiwari SK. Probiotics, prebiotics and synbiotics: Safe options for next-generation therapeutics. Appl Microbiol Biotechnol. 2022 Jan;106(2):505-521. doi: 10.1007/s00253-021-11646-8. Epub 2022 Jan 11. PMID 35015145
- [Background] Kobyliak N, Abenavoli L, Mykhalchyshyn G, Kononenko L, Boccuto L, Kyriienko D, Dynnyk O. A Multi-strain Probiotic Reduces the Fatty Liver Index, Cytokines and Aminotransferase levels in NAFLD Patients: Evidence from a Randomized Clinical Trial. J Gastrointestin Liver Dis. 2018 Mar;27(1):41-49. doi: 10.15403/jgld.2014.1121.271.kby. PMID 29557414
- [Background] Abhari K, Saadati S, Yari Z, Hosseini H, Hedayati M, Abhari S, Alavian SM, Hekmatdoost A. The effects of Bacillus coagulans supplementation in patients with non-alcoholic fatty liver disease: A randomized, placebo-controlled, clinical trial. Clin Nutr ESPEN. 2020 Oct;39:53-60. doi: 10.1016/j.clnesp.2020.06.020. Epub 2020 Jul 24. PMID 32859329
- [Background] Manzhalii E, Virchenko O, Falalyeyeva T, Beregova T, Stremmel W. Treatment efficacy of a probiotic preparation for non-alcoholic steatohepatitis: A pilot trial. J Dig Dis. 2017 Dec;18(12):698-703. doi: 10.1111/1751-2980.12561. PMID 29148175
- [Background] Chong CYL, Orr D, Plank LD, Vatanen T, O'Sullivan JM, Murphy R. Randomised Double-Blind Placebo-Controlled Trial of Inulin with Metronidazole in Non-Alcoholic Fatty Liver Disease (NAFLD). Nutrients. 2020 Mar 27;12(4):937. doi: 10.3390/nu12040937. PMID 32230987
- [Background] Behrouz V, Aryaeian N, Zahedi MJ, Jazayeri S. Effects of probiotic and prebiotic supplementation on metabolic parameters, liver aminotransferases, and systemic inflammation in nonalcoholic fatty liver disease: A randomized clinical trial. J Food Sci. 2020 Oct;85(10):3611-3617. doi: 10.1111/1750-3841.15367. Epub 2020 Sep 4. PMID 32885440
- [Background] Bakhshimoghaddam F, Shateri K, Sina M, Hashemian M, Alizadeh M. Daily Consumption of Synbiotic Yogurt Decreases Liver Steatosis in Patients with Nonalcoholic Fatty Liver Disease: A Randomized Controlled Clinical Trial. J Nutr. 2018 Aug 1;148(8):1276-1284. doi: 10.1093/jn/nxy088. PMID 29931231
- [Background] Ahn SB, Jun DW, Kang BK, Lim JH, Lim S, Chung MJ. Randomized, Double-blind, Placebo-controlled Study of a Multispecies Probiotic Mixture in Nonalcoholic Fatty Liver Disease. Sci Rep. 2019 Apr 5;9(1):5688. doi: 10.1038/s41598-019-42059-3. PMID 30952918
- [Background] Chen Y, Feng R, Yang X, Dai J, Huang M, Ji X, Li Y, Okekunle AP, Gao G, Onwuka JU, Pang X, Wang C, Li C, Li Y, Sun C. Yogurt improves insulin resistance and liver fat in obese women with nonalcoholic fatty liver disease and metabolic syndrome: a randomized controlled trial. Am J Clin Nutr. 2019 Jun 1;109(6):1611-1619. doi: 10.1093/ajcn/nqy358. PMID 31136662